CLINICAL TRIAL: NCT03772665
Title: A Phase 3 Multicenter, Randomized, Double-Masked Study Comparing the Efficacy and Safety of Emixustat Hydrochloride With Placebo for the Treatment of Macular Atrophy Secondary to Stargardt Disease
Brief Title: Safety and Efficacy of Emixustat in Stargardt Disease
Acronym: SeaSTAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kubota Vision Inc. (Industry)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4429-301; R01FD006849 (FDA)
Record Dates: First submitted 2018-11-30; First posted 2018-12-11 (Actual); Results first posted 2023-08-03 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Stargardt Disease
Keywords: Stargardt Disease; STGD; ABCA4
MeSH Terms: conditions — Stargardt Disease | interventions — emixustat

STUDY DESIGN:
Intervention Model Description: This is a multicenter, randomized, double-masked, placebo-controlled study to evaluate the efficacy and safety of emixustat compared to placebo in subjects who have Macular Atrophy secondary to Stargardt disease.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Emixustat (Experimental): 10 mg
  Interventions: Drug: Emixustat
- Placebo (Placebo Comparator): Includes identical tablets with only inactive ingredients (0 mg).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Emixustat — Once daily oral tablet taken for 24 months
  Other Names: emixustat hydrochloride
  Arms: Emixustat
Drug: Placebo — Once daily oral tablet taken for 24 months
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if emixustat hydrochloride reduces the rate of progression of macular atrophy compared to placebo in subjects with Stargardt disease.

Funding Source -- FDA OOPD

DETAILED DESCRIPTION:
Stargardt disease is a rare, inherited degenerative disease of the retina affecting approximately 1 in 8000 to 10 000 people and is the most common type of hereditary macular dystrophy. There are no approved treatments for STGD. This disease is characterized by an excessive accumulation of lipofuscin at the level of the retinal pigment epithelium (RPE). Lipofuscin is made of lipids, proteins, and toxic bis retinoids (such as N retinylidene N retinylethanolamine [A2E]). Accumulation of the toxic bis retinoids found in lipofuscin is thought to cause RPE cell dysfunction and eventual apoptosis, resulting in photoreceptor death and loss of vision.

Stargardt disease has several sub types, where autosomal recessive STGD (STGD1) accounts for the majority (>95%) of all cases. STGD1 is typically diagnosed in the first 3 decades of life and is caused by mutations of the adenosine triphosphate binding cassette subfamily A member 4 (ABCA4) gene. The ABCA4 gene product transports N retinylidene phosphatidylethanolamine (a precursor of toxic bis retinoids) from the lumen side of photoreceptor disc membranes to the cytoplasmic side where the retinal is hydrolyzed from phosphatidylethanolamine. Mutations of the ABCA4 gene result in accumulation of this precursor in disc membranes that are eventually phagocytized by RPE cells, where the precursors are converted into toxic bis retinoids such as A2E. In addition to being a precursor to A2E, all trans retinal has also been implicated in the pathogenesis of STGD through its role in light-mediated toxicity.

Emixustat hydrochloride (emixustat) has been developed by Acucela Inc. for retinal diseases including Stargardt disease (STGD). Emixustat is a potent inhibitor of RPE65 isomerization activity and reduces visual chromophore (11 cis retinal) production in a dose-dependent and reversible manner. Because 11 cis-retinal and its photoproduct (all trans retinal) are substrates for biosynthesis of retinoid toxins (eg, A2E), chronic treatment with emixustat retards the rate at which these toxins accumulate.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of macular atrophy secondary to Stargardt disease (STGD)
* Macular atrophy measured to fall within a defined size range
* Two mutations of the ABCA4 gene. If only one mutation, a typical STGD appearance of the retina.
* Visual acuity in the study eye of at least 20/320

Exclusion Criteria:

* Macular atrophy secondary to a disease other than STGD
* Mutations of genes, other than ABCA4, that are associated with retinal degeneration
* Surgery in the study eye in the past 3 months
* Prior participation in a gene therapy or stem cell clinical trial for STGD
* Recent participation in a clinical trial for STGD evaluating a complement inhibitor or vitamin A derivative
* Use of certain medications in the past 4 weeks that might interfere with emixustat
* An abnormal electrocardiogram (ECG)
* Certain abnormalities on laboratory blood testing
* Female subjects who are pregnant or nursing

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Gregory, MD, Study Director — VP of Clinical Development, Acucela
Locations (29):
- United States (11):
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - UCSF Dept. of Ophthalmology, San Francisco, California
  - Emory University, Atlanta, Georgia
  - The Wilmer Eye Institute Johns Hopkins University, Baltimore, Maryland
  - University of Michigan Kellogg Eye Center, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Duke Eye Center, Durham, North Carolina
  - Casey Eye Institute - OHSU, Portland, Oregon
  - Retina Foundation of the Southwest, Dallas, Texas
  - University of Utah John Moran Eye Center, Salt Lake City, Utah
  - Medical College of Wisconsin-Eye Institute, Milwaukee, Wisconsin
- Brazil (2):
  - Santa Casa de Misericórdia de Belo Horizonte, Belo Horizonte, Minas Gerais
  - Hospital Sao Paulo, São Paulo
- The Hospital for Sick Children, Toronto, Ontario, Canada
- Rigshospitalet-Glostrup, Glostrup Municipality, Capital Region, Denmark
- France (2):
  - Service D'Ophtalmologie Chi Creteil, Créteil, Île-de-France Region
  - CHNO Quinze-Vingts - CIC, Paris, Île-de-France Region
- Germany (2):
  - Universitätsklinikum Tübingen, Department für Augenheilkunde, Tübingen, Baden-Wurttemberg
  - Universitäts-Augenklinik Bonn, Bonn
- Italy (5):
  - AOU Università della Campania Luigi Vanvitelli, Naples, Campania
  - Università Cattolica del Sacro Cuore - Fondazione Policlinico Gemelli, Rome, Lazio
  - IRCCS Ospedale San Raffaele, Milan, Lombardy
  - UOC Oculistica Asst Fatebene Pratelli Sacco Universita delgi Studi di Milano, Milan, Lombardy
  - SODC di Oculistica AOU Careggi, Florence, Tuscany
- Radboud University Medical Center, Nijmegen, Gelderland, Netherlands
- Pretoria Eye Institute, Pretoria, Gauteng, South Africa
- Fundacion Jimenez Diaz University Hospital, Madrid, Spain
- United Kingdom (2):
  - Oxford Eye Hospital,Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire
  - Moorfields Eye Hospital NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Emixustat | Placebo
Started | 128 | 66
Completed | 127 | 66
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: ITT
Groups:
- Total: Total of all reporting groups
Arm/Group | Emixustat | Placebo | Total
Number analyzed (Participants) | 128 | 66 | 194
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 2 | 7
  Between 18 and 65 years | 122 | 64 | 186
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (15.03) | 43.0 (14.07) | 43.6 (14.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 29 | 88
  Male | 69 | 37 | 106
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 3 | 2 | 5
  Netherlands | 3 | 2 | 5
  United States | 34 | 19 | 53
  Brazil | 20 | 9 | 29
  Denmark | 6 | 4 | 10
  Italy | 24 | 9 | 33
  South Africa | 11 | 7 | 18
  United Kingdom | 6 | 3 | 9
  France | 8 | 4 | 12
  Germany | 8 | 5 | 13
  Spain | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Mean Rate of Change in Total Area of Macular Atrophy, as Measured by Fundus Autofluorescence (FAF)
Description: Mean rate of change in total area of macular atrophy, as measured by fundus autofluorescence (FAF)
Time Frame: 24 months
Population: ITT
Measure: Mean (Standard Error); unit: Rate of change from BL (mm^2/yr)
Arm/Group | Emixustat | Placebo
Number analyzed (Participants) | 128 | 66
Rate of change from BL (mm^2/yr) | 1.280 (0.0783) | 1.309 (0.1002)

ADVERSE EVENTS:
Time Frame: 24 months
Description: MedDRA version 25.0
Arm/Group | Emixustat | Placebo
All-Cause Mortality (participants affected / at risk) | 0/127 | 0/66
Serious Adverse Events (participants affected / at risk) | 9/127 | 2/66
Other Adverse Events (participants affected / at risk) | 1/127 | 0/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Emixustat (N=127) | Placebo (N=66)
agina pectoris (Cardiac disorders) | 1 (1) | 1 (1)
atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Infections and infestations (Infections and infestations) | 1 (1) | 1 (1)
Visual disorder (Eye disorders) | 1 (1) | 0 (0)
Injury, posioning and procedural (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nervous system disorder (Nervous system disorders) | 1 (1) | 0 (0)
Vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Emixustat (N=127) | Placebo (N=66)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-21): https://cdn.clinicaltrials.gov/large-docs/65/NCT03772665/Prot_SAP_000.pdf